CLINICAL TRIAL: NCT01365403
Title: A SINGLE CENTER, OPEN LABEL, FIXED SEQUENCE, TWO-PERIOD STUDY TO INVESTIGATE THE EFFECT OF MULTIPLE DOSE CARBAMAZEPINE ON SINGLE DOSE PHARMACOKINETICS OF RO4917838 IN HEALTHY MALE VOLUNTEERS
Brief Title: A Study on The Effect of Multiple Dose Carbamazepine on Single Dose Pharmacokinetics of RO4917838 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: BP25263
Record Dates: First submitted 2011-05-20; First posted 2011-06-03 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Carbamazepine

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: RO4917838; Drug: carbamazepine

INTERVENTIONS:
Drug: RO4917838 — Single oral dose, Day 1 of study period 1 and Day 16 of study period 2
Drug: carbamazepine — multiple oral doses, Days 1-24 of study period 2

SUMMARY:
This open-label, fixed sequence, two-period study will assess the effect of multiple dose carbamazepine on the single dose pharmacokinetics of RO4917838. Subjects will receive a single oral dose of RO4917838 on Day 1 of the 12-day study period 1 and, after a washout of 3-6 weeks, in study period 2 carbamazepine orally daily on Days 1-24 with a single oral dose of RO4917838 on Day 16.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy male volunteers, 18-65 years of age inclusive
* Body mass index (BMI) 18-30 kg/m2 inclusive

Exclusion Criteria:

* History or presence of any disorder or condition that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the investigator
* History of any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, allergic, dermatologic, hematologic, neurologic or psychiatric disease, or cancer
* Any confirmed significant allergic reactions against any drug, or multiple allergies in the judgment of the investigator
* Native Asians or subjects with Asian racial origin

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Area under the concentraion-time curve/maximum concentration (AUC/Cmax) of single dose RO4917838 with multiple dose carbamazepine administration | approximately 4 weeks

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | up to 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Rennes, France